CLINICAL TRIAL: NCT00240851
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating Acetaminophen Extended Release Caplets (3900 mg/Day) in the Treatment of Post-Race Muscle Aching and Pain (Soreness)
Brief Title: An Effectiveness and Safety Study of Acetaminophen Extended Release Caplets in Treating Muscle Aches and Soreness That Occur After a Marathon Race
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002881
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Pain
Keywords: muscle ache; pain; soreness; acetaminophen
MeSH Terms: conditions — Pain; Myalgia

ARMS (1):
- 001 (Experimental): acetaminophen extended release
  Interventions: Drug: acetaminophen extended release

INTERVENTIONS:
Drug: acetaminophen extended release

SUMMARY:
The purpose of this study is to compare the effectiveness of acetaminophen extended release caplets to placebo in treating the muscle aching and pain (soreness) that occurs after a marathon.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to compare the effectiveness and safety of acetaminophen and placebo in treating muscle aching and pain (soreness) that occurs in subjects who complete a marathon. Subjects are randomized to receive acetaminophen extended release caplets, 3900 mg/day (two 650 mg caplets taken three times a day, for four days) or placebo (two placebo caplets taken three times a day, for four days). The primary measurement of efficacy is the average change from baseline in muscle soreness, on Day 1, the day of the marathon. Safety assessments consist of monitoring adverse events, and a physical examination at the screening visit, including vital signs, weight, a medical history review, and a urine pregnancy test for females of childbearing potential. The hypothesis of the study is that acetaminophen is more effective than placebo in the relief of post-race muscle aching and pain (soreness) score on the evening of the race. Two acetaminophen 650 mg extended release caplets, taken by mouth, three times a day over a four day period or two placebo caplets, taken by mouth, three times a day over a four day period.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to comply with the study schedule
* be able to swallow the study medication
* complete the marathon
* not take any analgesics after completing the marathon and before their eligibility to participate in the study has been determined
* rate their muscle soreness at least a 4, on a 0 - 10 point scale

Exclusion Criteria:

* Previous diagnosis of osteoarthritis
* currently have or have had a medical condition that may be relevant in one's eligibility to participate in the study
* known hypersensitivity to acetaminophen
* unable to understand or follow the instructions for the study
* taken any investigational medication within 30 days of the marathon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
The average change from baseline in muscle soreness on Day 1

SECONDARY OUTCOMES:
Average change from baseline in muscle soreness for both morning and evening assessments, combined and separately; Average ratings of interference with 1) sleep, 2) daily activity, and 3) ability to go for a run

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- See also: An Effectiveness and Safety Study of Acetaminophen Extended Release Caplets in Treating Muscle Aches and Soreness that Occur After a Marathon Race — http://download.veritasmedicine.com/PDF/CR002881_CSR.pdf